CLINICAL TRIAL: NCT03386682
Title: Evaluation of the Safety and Performance of SYMATESE AESTHETICS ESTYME® MATRIX Round and Anatomical Silicone Gel-Filled Breast Implants in the Breast Augmentation and Reconstruction - EMMIE Study
Brief Title: Evaluation of the Safety and Performance of ESTYME® MATRIX Round and Anatomical Breast Implants - EMMIE Study
Acronym: EMMIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Symatese Aesthetics (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol CLIN PMI-002
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Breast Augmentation; Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESTYME MATRIX (Experimental): Participants who meet the requirements for breast augmentation or breast reconstruction surgeries and have been implanted with one or two ESTYME® MATRIX Breast Implant(s)
  Interventions: Device: ESTYME® MATRIX Breast Implants

INTERVENTIONS:
Device: ESTYME® MATRIX Breast Implants — Breast implant surgery in breast reconstruction or breast augmentation

SUMMARY:
The study will evaluate the safety and performance of the ESTYME® MATRIX Round and Anatomical Silicone Gel-Filled Breast Implants in the breast augmentation and reconstruction.

DETAILED DESCRIPTION:
The study will evaluate the safety and performance of the ESTYME® MATRIX Round and Anatomical Silicone Gel-Filled Breast Implants in the breast augmentation and reconstruction at 3 months, 1 year and 2 years post-procedure

ELIGIBILITY:
Inclusion Criteria:

Patient will be included if all of the following criteria are met:

1. Subject of between 18 and 65 years old
2. Candidate eligible for :

   a. unilateral or bilateral breast augmentation i. general breast enlargement: cosmetic purposes, providing symmetry to opposite breast in case of unilateral surgery ii. surgical correction of various congenital or acquired anomalies such as amastia, aplasia, hypomastia, hypoplasia, asymmetries, Poland's syndrome, ptosis …

   b. or immediate or delayed unilateral or bilateral breast reconstruction (for cancer, trauma, surgical loss of breast)
3. Patient signs PIC (Patient Informed Consent) & willing to comply with the protocol assessments and visits follow up

Exclusion Criteria:

Patient will not be included if any of the following conditions exists:

1. Local or systemic infection or abscess anywhere in the body
2. Existing carcinoma or pre-carcinoma of the breast without treatment or mastectomy treatment without appropriate wash out period for chemotherapy at the surgeon discretion
3. Subject with previous tissue expansion
4. Diagnosis of active cancer of any type for augmentation procedure subject
5. Pregnant subject or intending to become pregnant within three (3) months of the implant procedure
6. Subject who had nursed within three (3) months of implant surgery, or still breastfeeding
7. Tissue characteristics determined clinically inadequate or unsuitable by the surgeon (i.e. tissue damage resulting from radiation, inadequate tissue or compromised vascularity, know complication wound healing)
8. Previously implanted subject with a silicone implant or History of failure following cosmetic augmentation or subcutaneous mastectomy
9. History of autoimmune disease such as but not limited to: lupus, scleroderma …
10. Any condition or treatment for any condition which, in the opinion of the physician, may constitute an unwarranted surgical risk (e.g. anaesthesia allergy, high consumption smoking subject …)
11. Anatomic or physiologic abnormality which could result to significant post-operative complications
12. History of sensitivity of foreign materials or known allergy to any component of the ESTYME® MATRIX Silicone Gel-Filled Breast Implant
13. Subject known for alcohol abuse/history
14. Underlying disease (HIV positive Subject, HF (heart Failure), renal insufficiency, diabetes, hypertension, …)
15. Subject with implanted metal or metal devices, history of claustrophobia, or other condition that would make a MRI scan prohibitive
16. Unwilling to undergo any further surgery for revision
17. Subject with willingness that are unrealistic/unreasonable with the risks involved with the surgical procedure
18. Participating into any other clinical study or had participated into a clinical study without appropriate wash out period at the surgeon discretion
19. Subject who has sociological, cultural or geographical factors which could interfere with evaluation or completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2021-04-12 (Estimated)

PRIMARY OUTCOMES:
Local complications | 3 months
  Evaluation of the safety 3 months post-implantation.
  Procedure-related adverse events/complications at 3 months post implant. Main foreseen complications: infection, haematoma, wound healing complication, fluid accumulation, early capsular contracture, rupture, extrusion.
Satisfaction of the patient and the surgeon | 3 months
  Evaluation of the performance, 3 months post-implantation
  Performance endpoint will be assessed by implant procedure success at 3 months defined as follows:
  * satisfactory procedure duration for the surgeon
  * satisfactory size of the incision for the surgeon
  * implant correct placement (absence of visible deformation of the gel, absence of rotation for anatomical implants)

SECONDARY OUTCOMES:
Local complications | 1 year and 2 years
  Evaluation of the safety, 1 year and two years post-implantation.
  Safety endpoint: incidence of all Adverse Events (AE)/Serious Adverse Events (SAEs) @ 1 year and two years post procedure
Satisfaction of the patient and the surgeon | 1 year and 2 years
  Performance endpoints are as follows:
  * global surgeon satisfaction post-procedure assessed by the usability of the device during the procedure (current implant procedure): surgeon comfort level for the insertion/implantation of the prosthesis,
  * global patient and surgeon satisfaction @ 1 year and 2 years post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: EMMANUEL DELAY, MD, Principal Investigator — Clinique Charcot
Locations (8):
- France (8):
  - Centre F.X. Michelet Chu Bordeaux, Bordeaux
  - Chu Pasteur, Nice
  - Clinique des Champs Elysées, Paris
  - Clinique BIZET, Paris
  - Institut du Sein, Paris
  - Hopital Tenon, Paris
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No